CLINICAL TRIAL: NCT00225368
Title: Long Term Effects of Insecticide Treated Bednets on the Morbidity and Mortality Caused by Malaria and on the Overall Mortality in Young Children of a Rural Population in Burkina Faso
Brief Title: Effects of Insecticide Treated Bednets on Child Morbidity and Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SFB 544 D4(1)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2005-09

CONDITIONS: Malaria; All-cause Mortality
Keywords: Malaria; All-cause mortality; Africa; Burkina Faso
MeSH Terms: conditions — Malaria | interventions — Insecticide-Treated Bednets

INTERVENTIONS:
Device: Insecticide treated bednets

SUMMARY:
Insecticide-impregnated bed nets and curtains (ITN) have been shown to be effective against malaria. However, given that most ITN studies were of limited length, researchers have postulated the hypothesis that in areas of intense malaria transmission and due to possible interactions with immunity development, ITN interventions may cause no effect at all or even a long-term increase in malaria morbidity and mortality.

The overall objective of the trial is to analyse the long-term effects of ITN on child morbidity and mortality in an area of intense malaria transmission. The specific objective is to analyse if there is a difference in the rates of malaria morbidity and mortality as well as in all-cause mortality in children being protected with ITNs from birth compared to children protected with ITNs from age 6 months onwards.

The study is conducted in the Nouna Health District, in Burkina Faso, and specifically in a sub-portion of the District under demographic surveillance since 1999. The sub-portion of the District under demographic surveillance includes a total population of 70 000 individuals, distributed in 42 villages and in the town of Nouna. The region is a dry Savannah characterised by high levels of malaria transmission.

The study design entails a prospective community-based trial, with newborn children being identified at the village level and then individually randomised to receive either intervention A or intervention B. Intervention A is defined as ITN protection from age 0 to 59 months (i.e. protection from birth). Intervention B is defined as ITN protection from age 6 to 59 months (i.e. protection from 6 months onwards). Enrollment in the study cohort in continued until the sample size is reached (n = 2 600, 1 300 group A and 1 300 group B).

Detailed data on morbidity is collected through means of a prospective follow up on a sub-sample of 420 children from 6 sentinel villages (210 from group A and 210 from group B). These 420 children are visited daily by field workers who measure their temperature. In case of fever, field workers take a blood sample through finger prick to be analysed for malaria parasitaemia. Treatment free of charge is organised for all children in this subsample. In addition, these children are visited twice a year for the collection of clinical (malaria episodes, anaemia) and parasitological (rates of malaria parasitaemia, parasite density) parameters. Data collection on this subsample of children is meant to last from June 2000 to December 2003. For study purposes, falciparum malaria is defined as 37.5 C or more plus at least 5 000 parasites per micro-litre.

All-cause mortality in the overall study sample (2 600 children) are ascertained through means of a demographic surveillance system (DSS), which regularly monitors deaths (as well as births and migration) in the region. The causes of death are identified through means of verbal autopsy. All children enrolled in the study are followed up through means of the DSS from birth up to 5 years of age.

The primary study outcome will be the five-year all-cause mortality in the total number of children enrolled in the study (2 600). Secondary outcomes will be the study of malaria-specific mortality, clinical parameters, and parasitological parameters in a sub-sample of the study cohort (420).

ELIGIBILITY:
Inclusion Criteria:

* Recruitment within two weeks from birth
* Being permanent resident in study village

Exclusion Criteria:

* Recruitment after two weeks from birth con
* Not being permanent resident in study village

Ages: 1 Day to 15 Days | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Mueller, MD, PhD, Principal Investigator — Heidelberg University
Locations (1):
- Nouna Health Research Centre, Nouna, Burkina Faso

REFERENCES:
- [Background] Muller O, Frey C, Traore C, Kouyate B. Retreatment of long-lasting insecticide-treated mosquito nets under field conditions in rural Burkina Faso. J Trop Pediatr. 2004 Dec;50(6):380-1. doi: 10.1093/tropej/50.6.380. No abstract available. PMID 15537731
- [Background] Muller O, Jahn A. Expanding insecticide-treated mosquito net coverage in Africa: tradeoffs between public and commercial strategies. Trop Med Int Health. 2003 Oct;8(10):853-6. doi: 10.1046/j.1365-3156.2003.01119.x. No abstract available. PMID 14516294
- [Background] Muller O, Ido K, Traore C. Evaluation of a prototype long-lasting insecticide-treated mosquito net under field conditions in rural Burkina Faso. Trans R Soc Trop Med Hyg. 2002 Sep-Oct;96(5):483-4. doi: 10.1016/s0035-9203(02)90411-6. PMID 12474472
- [Background] Okrah J, Traore C, Pale A, Sommerfeld J, Muller O. Community factors associated with malaria prevention by mosquito nets: an exploratory study in rural Burkina Faso. Trop Med Int Health. 2002 Mar;7(3):240-8. doi: 10.1046/j.1365-3156.2002.00856.x. PMID 11903986